CLINICAL TRIAL: NCT05779787
Title: COronary Re-EngageMent aFter RandOm NavitoR Alignment (COMFORT STUDY)
Acronym: COMFORT
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D001024
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAVR performed with commissural alignment technique (Aligned Group): Patients with severe aortic stenosis undergoing TAVR procedure performed with commissural alignment technique. We consider in this groups only the Accurate and Accurate Neo 2 Valve which are the first choice due to the best stent frames position predictability with this technique
  Interventions: Procedure: TAVR Aligned; Procedure: TAVR Random
- TAVR performed with random implantation of Navitor valve (Random Group): Patients with severe aortic stenosis undergoing TAVR procedure performed with random implantation of Navitor Valve
  Interventions: Procedure: TAVR Aligned; Procedure: TAVR Random

INTERVENTIONS:
Procedure: TAVR Aligned — Investigate the feasibility of coronary re-engagement after commissural alignment technique in terms of success rate (%) and procedure complexity taking into account radiations, time and contrast used.
Procedure: TAVR Random — TAVR Random Feasibility comparison of coronary re-engagement between the randomly implanted Navitor valve (unaligned) and the others implanted with the commissural alignment technique in terms of success rate (%) and complexity of the procedure, taking into account radiation, time and contrast used

SUMMARY:
Whereas PCI before TAVR was previously recommended despite its uncertain prognostic role, recent data underline the possibility of a postponed coronary intervention using a commissural alignment technique. This approach allows easy coronary re-engagement through the valve stent frame with a trade off paid of procedure complexity.

Considering the prevalence of coronary artery disease (CAD) and the increasing percentage of younger patients treated with TAVI, investigate whether a simpler procedure with random implantation of Navitor valve is not inferior in terms of coronary re-access, is required The key point of the project will be the evaluation of the feasibility of coronary re-engagement after a Navitor valve randomly implanted.

DETAILED DESCRIPTION:
Transcatheter Aortic Valve Implantation (TAVI) is recommended by European and American guidelines to treat patients with aortic stenosis regardless of procedural risk (1, 2). In the last decades the increasing percentage of younger patients treated with TAVI, reflect the extensive indications in lower risk setting, highlighting the importance of easy coronary re-engagement after valve implantation. Considering the prevalence and the progression of a pre-existing coronary artery disease (CAD), the timing of coronary intervention should be accurate selected (3) addressing the percentage of unplanned percutaneous coronary intervention (PCI) after TAVI (4). In fact, while PCI before TAVR was previously recommend despite the uncertain prognostic role (5), recent data remarks the possibility of a postponed coronary intervention using a commissural alignment technique (6) that allows a predictable stent frame position in the sinus of Valsalva (7). Moreover, following the emerging concept of easy re-access, only a few types of prostheses have been shown to have an high degree of stent position predictability after implantation, leading to a limited option in terms of prosthesis choice. Furthermore, to achieve the best results with commissural alignment technique, accurate procedure planning and operator's expertise are required in order to properly manage the valve specific orientation in the aorta with consequent increase in time, radiation and procedure complexity.

However, geometry of the stent frame (height and size) and the anatomical characteristics of patients have to be enlisted as contributory factors to difficult coronary re-engagement and need to be evaluate in order to establish the feasibility of the re-access after TAVR.

The investigators' findings could provide data regarding the non-inferiority rate of coronary cannulation after a simpler procedure with Navitor implantation without alignment technique. Due to these results, the valves portfolio available in patients with coronary artery disease that needed PCI after TAVR, could be larger and various allowing the best protheses choice according to the patient's anatomy and operator's expertise. Finally, knowing the predictors of difficult re-engagement for both types of valves, regardless of implantation technique, could be interesting for an even more valve tailored approach.

The purpose of this study is to investigate the feasibility of coronary re-engagement after randomly (not aligned) Navitor implantation, as already perform in current clinical practice, due to a lower predictable orientation of this type of valve.

ELIGIBILITY:
Patients to be included in this registry should have all the following criteria:

1. Severe, symptomatic aortic stenosis with an indication to TAVI

Exclusion criteria and definition

Patients excluded in this registry should have all the following criteria:

1. Valve in Valve procedure
2. Hemodynamical instability
3. TAVR performed from other access (not femoral)
4. No-CT Planned TAVR
5. TAVR performed with Chimney Technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with severe aortic stenosis diagnosed according to ESC guidelines, undergoing transcatheters aortic valve replacement with Navitor valve randomly implanted or Acurate Neo with commisural alignment technique
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Coronary re-access after TAVR procedure | During procedure
  Re-engagement of LMCA and RCA after valve implantation is defined as selective cannulation and subsequent selective angiography. All others type of re-engagement will be classify as "non selective". We will stratify also the modality of re-cannulation in relation to the position of the valves' stent struts as "above", "across" and "behind".

SECONDARY OUTCOMES:
Total Implant Time | During procedure
  Total time required for valve implantation. We count the time from the alignment in the aorta to the end of valve opening (Alignment Fluoroscopy time + Implantation Fluoroscopy time).
Total Implant Fluoroscopy Time | During procedure
  Total Fluoroscopy time required for valve implantation. We count the time from the alignment in the aorta to the end of valve opening (Alignment time + Implantation time).
Total Implant Radiations | During procedure
  Total Radiations required for valve implantation. We count the radiations used from the alignment in the aorta to the end of valve opening (Alignment time + Implantation time).
Total Implant Contrast | During procedure
  Total Contrast required for valve implantation
Alignment Radiation | During procedure
  Radiation required for commissural alignment
Alignment Fluoroscopy Time | During procedure
  Fluoroscopy time required for commissural alignment
Implant Radiation | During procedure
  Radiation required for valve implantation
Implant Fluoroscopy Time | During procedure
  Fluoroscopy time required for valve implantation
Implant Contrast | During procedure
  Contrast required for valve implantation
Re-Engagement Radiation | During procedure
  Radiation required for re-engagement
Re-Engagement Fluoroscopy Time | During procedure
  Fluoroscopy time required for coronary re-engagement
Re-Engagement Contrast used | During procedure
  Contrast required for coronary re-engagement
Re-Engagement Time | During procedure
  Time required for coronary re-engagement

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided